CLINICAL TRIAL: NCT06275191
Title: Alternatives to Dental Opioid Prescribing After Tooth Extraction
Acronym: ADOPT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Oyler (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor-Investigator, Douglas Oyler, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 80758; 1UG3DE032621-01 (NIH); 4UH3DE032621-02 (NIH)
Record Dates: First submitted 2024-02-03; First posted 2024-02-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Analgesics, Opioid; Acute Pain; Tooth Extraction; Adolescent; Acetaminophen; Ibuprofen
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Who Masked: Participant, Investigator
Masking Description: Blinding to the intervention is not possible in this study, as the intervention requires provider engagement. Provider participants and any clinic personnel will be blinded to the allocation sequence, and those not yet receiving the intervention will not be aware of the time at which they will have the intervention implemented. The study biostatistician will be aware of the allocation sequence.
  At the beginning of each period, the study biostatistician will inform the research coordinator, project manager, academic detailing pharmacist, and PIs which cluster will be transitioning to the intervention condition next. This information will be used to facilitate scheduling academic detailing visits and coordinate blister pack and patient instructions material assembly. The clinic will be informed of their allocation during Visit 4 to facilitate scheduling academic detailing visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention condition (Experimental): 1. Academic detailing (45 to 60-minute session), plus
  2. Provision of standardized patient post-extraction instructions for distribution, plus
  3. Provision of blister-packaged acetaminophen and ibuprofen at recommended standard doses for distribution to to adolescent/young adult patients after tooth extraction in the course of clinical practice
  Interventions: Behavioral: Multicomponent intervention
- Control condition (Active Comparator): Usual practice
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Multicomponent intervention — The multicomponent intervention consists of (1) a single 45-60-minute academic detailing session with provider participants, plus (2) provision of patient post-extraction instruction materials and (3) provision of blister-packaged acetaminophen and ibuprofen for distribution to adolescent/young adult patients after tooth extraction in the course of clinical practice
  Arms: Intervention condition
Other: Usual care — No intervention.
  Arms: Control condition

SUMMARY:
The goal of this clinical trial is to test a three-item intervention in oral surgeons who remove teeth. The main questions it aims to answer are:

* Can the intervention reduce opioid prescriptions to adolescents and young adults after tooth removal?
* Do oral surgeons' beliefs about the intervention and opioid prescribing change?
* Do patients that report using opioids after tooth removal have different experiences than patients that do not?

Oral surgeon participants will:

* Attend a 1-hour education session with a trained pharmacist
* Receive patient instructions and blister packs of pain medicine to give to patients
* Complete 2 surveys about feasibility and appropriateness

Patient participants will complete a survey about pain and medication use after having a tooth removed.

Researchers will compare the intervention to usual care to see if it reduces opioid prescribing.

DETAILED DESCRIPTION:
Although use of nonsteroidal antiinflammatory drugs and acetaminophen is recommended first-line by the American Dental Association and American Association of Oral and Maxillofacial Surgeons, dentists and oral surgeons are leading prescribers of opioids to adolescents and young adults (AYA), who are at high risk for developing problematic opioid use after an initial exposure. This multi-site, stepped wedge cluster-randomized trial will assess whether a multicomponent behavioral intervention can influence opioid prescribing behavior among dentists and oral surgeons compared to usual practice. Across up to 12 clinical practices (clusters), up to 33 dentists and oral surgeons (provider participants) who perform tooth extractions for individuals 12-25 years old will be enrolled. After enrollment, all provider participants will receive the intervention at a time based on the sequence to which their cluster is randomized. The intervention consists of academic detailing plus provision of standardized patient post-extraction instructions and blister packs of acetaminophen (APAP) and ibuprofen for dispensing. Provider participants will dispense the blister packs and distribute the patient instructions at their discretion to AYA undergoing tooth extraction, with or without additional analgesics (e.g., opioids). The primary outcome is a binary, patient-level indicator of electronic post-extraction opioid prescription. Data for the primary outcome will be collected from the provider participant's electronic health records quarterly throughout the study. Provider participants will complete a survey before and approximately 3 months after transitioning into the intervention condition to assess implementation outcomes. AYA patients undergoing tooth extraction will be offered a survey to assess pain control and satisfaction with pain management in the week after their extraction. Primary analyses will use generalized estimating equations to compare the binary patient-level indicator of being prescribed a post-extraction opioid in the intervention condition compared to the control condition (i.e., usual practice). Analyses will adjust for patient-level factors (e.g., sex, number of teeth extracted, etc.). Secondary analyses will assess provider participants' perceptions of feasibility and appropriateness of the intervention, and patient-reported pain control and satisfaction with pain management.

ELIGIBILITY:
Inclusion Criteria (Provider):

* Actively U.S. licensed dentist or oral surgeon practicing at a participating cluster. Participating clinics were finalized prior to the beginning of the study based on the following criteria: (1) perform tooth extractions on at least 70 AYA patients during a 5-month screening period from July 1, 2022 through November 30, 2022 and (2) electronically prescribe opioids to at least 30% of AYA patients who underwent extraction during the screening period. Additionally, each participating cluster signed a data use agreement (DUA) for sharing electronic health record data, can provide the necessary electronic health record data, and agreed to comply with study procedures and be available for the duration of the study.
* Provide a signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.

Inclusion Criteria (Patient):

* Undergoes any tooth extraction at a participating cluster during the study (intervention condition, transition period, or control condition) between 6-10 days earlier.
* Age 12-25 at the time of tooth extraction.
* Reads and acknowledges survey cover letter in lieu of a full consent/assent process.
* Can access the electronic survey using an internet-capable device.

Exclusion Criteria:

* There are no other exclusion criteria for clusters or provider/patient participants that meet all inclusion criteria.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38159 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Odds of post-extraction opioid prescription to adolescent/young adults after tooth extraction | Same calendar date as dental extraction. Electronic health records will be extracted for the duration of the 4-year study period.
  The primary outcome is a patient-level binary indicator for being prescribed an opioid. The value for this outcome variable is equal to 1 if the patient is prescribed an opioid, whereas this variable takes on a value of 0 if this patient is not prescribed an opioid. Opioid prescription will be defined as an electronic order (from the electronic health record) for an opioid analgesic (e.g., hydrocodone, oxycodone, tramadol, morphine, fentanyl, etc.) on the same calendar date as the tooth extraction appointment.

SECONDARY OUTCOMES:
(Change in) intervention feasibility | Pre-surveys will be conducted during the calendar month preceding the transition to the intervention condition (i.e., within 60 days). Post-surveys will be conducted during the 3rd month of the intervention condition (i.e., within 120 days).
  Survey response. 5-point Likert-type questions (from 1-completely disagree to 5-completely agree) regarding feasibility of distributing blister packs and patient post-extraction materials. Selection of the top 2 choices (completely agree or agree) from the scale is considered as agreement with the statement.
(Change in) intervention appropriateness | Pre-surveys will be conducted during the calendar month preceding the transition to the intervention condition (i.e., within 60 days). Post-surveys will be conducted during the 3rd month of the intervention condition (i.e., within 120 days).
  Survey response. 5-point Likert-type questions (from 1-completely disagree to 5-completely agree) regarding appropriateness of distributing blister packs and patient post-extraction materials. Selection of the top 2 choices (completely agree or agree) from the scale is considered as agreement with the statement.
(Change in) opioid prescribing feasibility | Pre-surveys will be conducted during the calendar month preceding the transition to the intervention condition (i.e., within 60 days). Post-surveys will be conducted during the 3rd month of the intervention condition (i.e., within 120 days).
  Survey response. 5-point Likert-type questions (from 1-completely disagree to 5-completely agree) regarding feasibility of reducing opioid prescription. Selection of the top 2 choices (completely agree or agree) from the scale is considered as agreement with the statement.
(Change in) opioid prescribing appropriateness | Pre-surveys will be conducted during the calendar month preceding the transition to the intervention condition (i.e., within 60 days). Post-surveys will be conducted during the 3rd month of the intervention condition (i.e., within 120 days).
  Survey response. 5-point Likert-type questions (from 1-completely disagree to 5-completely agree) regarding appropriateness of reducing opioid prescription. Selection of the top 2 choices (completely agree or agree) from the scale is considered as agreement with the statement.
Self-reported pain | within 10 days of tooth extraction
  Patient survey, 3 items from Brief Pain Inventory (worst, least, average pain) based on self-reported opioid use. Each item uses an 11-point Visual Rating Scale from 0-no pain to 10-worst possible pain.
Self-reported pain interference | within 10 days of tooth extraction
  Patient survey, NIH PROMIS Pediatric Short Form v1.0-Pain Interference 8a (age < 18) or NIH PROMIS Adult Short Form v1.0-Pain Interference 6b (18+) based on self-reported opioid use. NIH PROMIS Pediatric Short Form t-scores range from 34.0 to 78.0, with higher scores indicating greater interference. NIH PROMIS Adult Short Form t scores range from 41.0 to 78.3, with higher scores indicating greater interference.
Self-reported pain satisfaction | within 10 days of tooth extraction
  Patient survey, 5-point Likert-type question (from 1-very unhappy to 5-very happy) regarding overall satisfaction with pain management based on self-reported opioid use. Selection of the top 2 choices (very happy or happy) from the scale is considered as satisfaction with overall pain management.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Oyler, PharmD, Principal Investigator — University of Kentucky; Marcia V Rojas Ramirez, DDS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oyler DR, Rojas-Ramirez MV, Nakamura A, Quesinberry D, Miller CS. Dental opioid prescription patterns in academic and community settings. J Public Health Dent. 2023 Jun;83(2):200-206. doi: 10.1111/jphd.12568. Epub 2023 Mar 11. PMID 36905202
- [Background] Oyler DR, Rojas-Ramirez MV, Nakamura A, Quesinberry D, Bernard P, Surratt H, Miller CS. Factors influencing opioid prescribing after tooth extraction. J Am Dent Assoc. 2022 Sep;153(9):868-877. doi: 10.1016/j.adaj.2022.05.001. Epub 2022 Jun 9. PMID 35691709
- [Background] Oyler DR, Miller CS. Patterns of opioid prescribing in an Appalachian college of dentistry. J Am Dent Assoc. 2021 Mar;152(3):209-214. doi: 10.1016/j.adaj.2020.12.002. PMID 33632410
- [Background] Oyler DR, Westgate PM, Walsh SL, Dolly Prothro J, Miller CS, Roberts MF, Freeman PR, Knudsen HK, Lang M, Dominguez-Fernandez E, Rojas-Ramirez MV. Alternatives to dental opioid prescribing after tooth extraction (ADOPT): protocol for a stepped wedge cluster randomized trial. BMC Oral Health. 2024 Apr 4;24(1):414. doi: 10.1186/s12903-024-04201-0. PMID 38575929